CLINICAL TRIAL: NCT02352792
Title: Randomized Phase II Study for Dose Escalation in Locally Advanced Head and Neck Squamous Cell Carcinomas Treated With Radiochemotherapy
Brief Title: Hypoxia-based Dose Escalation With Radiochemotherapy in Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.0
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Local control
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy (Active Comparator): Standard radiochemotherapy (70 Gy, 5-fluorouracil 600 mg/m2 d1-5, mitomycin C d1+36 or cisplatinum 40 mg/m2 weekly for 5 weeks)
  Interventions: Radiation: radiochemotherapy with 70 Gy
- dose escalation (Experimental): Standard plus 10% dose escalation to the hypoxic volume
  Interventions: Radiation: radiochemotherapy with 77 Gy

INTERVENTIONS:
Radiation: radiochemotherapy with 70 Gy
  Arms: Standard therapy
Radiation: radiochemotherapy with 77 Gy
  Arms: dose escalation

SUMMARY:
Patients with locally advanced suqamous cell carcinoma of the head and neck region receive a hypoxia scan either by magnetic resonance tomography, computed tomography or fluoromisonidazole (FMISO)-PET-CT. Patients presenting with hypoxia are randomized into standard therapy consisting of intensity modulated radiotherapy (IMRT) with 70 Gy plus either 5-fluorouracil/mitomycin C or cisplatinum (Arm A) or a dose escalation of 10% (77Gy) to the hypoxic volume applied via simultaneous integrated boost in addition to the standard treatment (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* histologically verified squamous cell carcinoma of the head and neck region stage III and IV eligible for primary radiochemotherapy
* measurabel disease by CT and/or MRT and/or FDG-PET-CT
* fit for chemotherapy
* no prior radiotherapy or major surgery in the head/neck region
* Karnofsky Index > 60%
* informed consent

Exclusion Criteria:

* uncontrolled secondary cancer
* distant metastases
* pregnancy
* expected malcompliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2017-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
time to local recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Welz, Dr. med., Principal Investigator — radiation oncology
Locations (1):
- Tuebingen university, radiation oncology, Tübingen, Baden-Wurttemberg, Germany